CLINICAL TRIAL: NCT03573440
Title: The Effects of Mindful Eating Education on Increasing Satiety Signals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Georgia Hodgkin, EdD, Associate Chair of Nutrition and Dietetics, Loma Linda University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 5180174
Record Dates: First submitted 2018-06-07; First posted 2018-06-29 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Mindfulness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no mindful eating education (No Intervention): * Subject will be asked to eat their meal with an investigator present.
  * They will inform the investigator verbally when they are feeling full.
  * After they have decided to end their meal, they will be asked to fill out a questionnaire
- mindful eating education (Experimental): * After receiving a brief education session on mindful eating, subject will be asked to eat their meal with an investigator present.
  * They will inform the investigator verbally when they are feeling full.
  * After they have decided to end their meal, they will be asked to fill out a questionnaire
  Interventions: Other: mindful education on eating

INTERVENTIONS:
Other: mindful education on eating — Mindful eating education material: mindful eating handout by move.va.gov. It includes topics such as: observe your body, do not judge yourself, notice your reaction to food and savor your food.
  Arms: mindful eating education

SUMMARY:
The purpose of this graduate student research study is to is to examine the effects of mindful eating education on increasing satiety signals.

Reasons for conducting the study: Add to the body of knowledge on the science of mindful eating.

DETAILED DESCRIPTION:
The procedures include:

Visit 1:

* The subject will be asked to meet the student investigators at the Loma Linda Student Pavilion, sign an informed consent form, sign in, and provide an email address and phone number.
* After the initial briefing, the subject will be asked to eat their meal with an investigator present.
* The subject will inform the investigator verbally when they are feeling full.
* After the subject decides to end their meal, the subject will be asked to fill out a questionnaire and be reminded to bring the same meal the following week.

Visit 2:

* The subject will be asked to meet the student investigators at the Loma Linda Student Pavilion with the same meal as the previous week.
* After receiving a brief education session, the subject will be asked to eat their meal with an investigator present.
* The subject must inform the investigator verbally when they are feeling full.
* After the subject has decided to end their meal, they will be asked to fill out a questionnaire and be reminded to meet the investigator at the same time the following week.

Visit 3:

* The subject will be asked to meet the student investigators at the Loma Linda Student Pavilion.
* The subject will be asked to complete a follow-up survey on the study.

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled at Loma Linda University
* pack or purchase their own lunch on a regular basis (willingness bring/buy the same lunch the following week)
* have a 1 hour or less lunch period.

Exclusion Criteria:

* skip breakfast
* have exercised within 2 hours of their lunch time
* smoke nicotine or marijuana
* have the condition of Type 1 or Type 2 diabetes
* have newly prescribed medications 2 weeks prior to testing.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change in satiety | change from baseline to one week
  The subject will be asked to verbally inform the investigator when they feel full. The investigator will be using a stopwatch to record when the subject has reached satiety.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Hodgkin, EdD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda Universtiy, Loma Linda, California, United States